CLINICAL TRIAL: NCT02103712
Title: Long Term Outcome of Hypospadias Repair: A Comparative Study
Brief Title: Long Term Outcome of Hypospadias Repair
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UR12/10496
Record Dates: First submitted 2013-11-20; First posted 2014-04-04 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypospadias
  Interventions: Other: Qualitative

INTERVENTIONS:
Other: Qualitative

SUMMARY:
Hypospadias is a common congenital abnormality of the penis which affects approximately 1 boy in 250. The opening of the urethra is located on the undersurface of the penis rather than the tip,the foreskin is deficient and there is curvature of the penile shaft in more severe cases. Although the most commonly practised corrective operation ( TIP procedure) gives generally good results, recently published evidence points to a possible long term risk of stenosis ( narrowing of the reconstructed urethra). This comparative study will combine clinical assessment with non invasive measurements of urinary flow to assess the functional outcome of a large series of patients who have undergone hypospadias surgery . The study is primarily designed to answer this question : does a modification of the standard operation which incorporates a skin graft into the reconstructed urethra lead to improved urinary flow and a decreased risk of stenosis? This has not been previously studied . The findings of our study could make an important contribution to improvements in the surgical treatment of boys born with hypospadias.

ELIGIBILITY:
Inclusion Criteria:

- 1 Patients with hypospadias who have been treated one of the following two surgical proceduresStandard Tubularised Incised Plate (TIP) operation (Group A) or Tubularised Incised Plate (TIP) procedure incorporating a free graft of preputial skin (in a layer of foreskin) into the urethral reconstruction (Group B ) 2 The study will be confined to primary operations. Patients in whom either of the techniques was used for a secondary or 'redo' procedure will be excluded from the study.

3 The study will be confined to boys over 3 years of age who are potty trained and able to pass urine for the non invasive flow rate test .

Exclusion Criteria:

- 1 Patients whose hypospadias was corrected using some technique other than 'standard' or 'grafted' TIP repair.

2 "Redo" cases 3 Boys under 3 years at the time of the study or patients who do not have full bladder control for some other reason.

Ages: 3 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with hypospadias
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Does a modification of the standard TIP hypospadias operation which incorporates a skin graft into the reconstructed urethra result in improved urinary flow and a (presumed)decrease in the long term risk of stenosis? | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom